CLINICAL TRIAL: NCT07372079
Title: Neoadjuvant Therapy for Early Triple-Negative Breast Cancer: A Response-Guided Approach Using Iparomlimab and Tuvonralimab Injection in Combination With Chemotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20251311
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Neoadjuvant Therapy; Immune Checkpoint Inhibitors; QL1706
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 Combination Therapy (Experimental): neoadjuvant QL1706 plus chemotherapy (four cycles of TP ± four cycles of AC).
  Interventions: Drug: QL1706 combined with Chemotherapy

INTERVENTIONS:
Drug: QL1706 combined with Chemotherapy — Participants receive QL1706 every 3 weeks (Q3W) + Albumin-bound paclitaxel every 3 weeks (Q3W) + Cisplatin (Q3W) x 4 cycles. After the four TP cycles, imaging and core biopsy will be performed. Patients who achieve radiologic complete response will proceed directly to surgery; those who do not will receive QL1706 Q3W + epirubicin Q3W + cyclophosphamide Q3W x 4 cycles as neoadjuvant therapy before surgery.

SUMMARY:
Iparomlimab and Tuvonralimab Injection (QL1706) is a bifunctional combination antibody targeting both programmed cell death protein 1 (PD-1) and cytotoxic T-lymphocyte antigen 4 (CTLA-4). This is a prospective clinical study that plans to enroll screened, eligible early-stage breast-cancer patients to receive neoadjuvant QL1706 plus chemotherapy (four cycles of TP ± four cycles of AC). After the four TP cycles, imaging and core biopsy will be performed. Patients who achieve radiologic complete response will proceed directly to surgery; those who do not will receive four additional AC cycles before surgery. A key feature is the incorporation of an response-guided neoadjuvant therapy（RGN）model to identify sensitive patients who can forgo anthracyclines, thereby reducing long-term cardiotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily join this study, sign the informed consent form, and demonstrate good compliance;
* Age: 18-75 years old (at the time of signing the informed consent form);
* ECOG PS score: 0-1; expected survival time exceeding 6 months;
* Patients with primary breast cancer confirmed by histopathological or cytological examination;
* Primary tumor diameter > 2 cm as measured by local standard assessment methods;
* Judged by the investigator to meet the American Joint Committee on Cancer (AJCC) 8th edition breast cancer TNM staging criteria as cT2-cT4, cN0-cN3, cM0, with locally advanced or early-stage, unilateral, and histologically confirmed invasive breast cancer;
* Histopathologically confirmed early-stage triple-negative invasive breast cancer as defined by the latest ASCO/CAP guidelines;
* At least one measurable lesion according to RECIST 1.1;
* The patient agrees to undergo breast cancer resection surgery when meeting the surgical criteria after neoadjuvant therapy;
* PD-L1 expression status is known;
* Major organ functions are in good condition;
* Female subjects of childbearing potential must have a negative serum pregnancy test within 3 days prior to the first dose. If a female subject of childbearing potential engages in sexual activity with a non-sterilized male partner, the subject must use acceptable and effective contraception from screening onward and agree to continue these precautions until 12 months after the last dose of the study drug; periodic abstinence and rhythm methods are not acceptable contraceptive methods.

Exclusion Criteria:

* Patients with stage IV metastatic breast cancer or other patients deemed by the investigator as unable to achieve curative surgical resection through neoadjuvant therapy;
* Patients with inflammatory breast cancer;
* Patients who have had or currently have other malignancies within the past 3 years. The following two conditions may be eligible: other malignancies treated with a single surgical procedure, achieving continuous 5-year disease-free survival (DFS); cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invading the basement membrane)];
* Breast cancer patients who have received antitumor therapies such as chemotherapy, endocrine therapy, or immune checkpoint inhibitors within the past 3 years, or who have undergone breast surgery (except diagnostic biopsy for primary breast cancer);
* Patients who have undergone major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of study treatment (except diagnostic biopsy for primary breast cancer);
* Presence of any active autoimmune disease or a history of autoimmune disease;
* Patients currently using immunosuppressants or systemic hormonal therapy for immunosuppressive purposes (at a dose >10 mg/day prednisone or equivalent steroids) and continuing such treatment within 2 weeks prior to enrollment;
* Allergy to any study drug or any component or excipient of the drug;
* Patients with concomitant diseases judged by the investigator as seriously endangering the subject's safety or affecting study completion, or those deemed unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04-05 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
tpCR（ypT0/is ypN0） | Up to approximately 27-30 weeks

SECONDARY OUTCOMES:
Radiologic complete response rate (iCR) | Up to approximately 27-30 weeks
epirubicin-cyclophosphamide regimen utilization rate | Up to approximately 16 weeks
Event-free Survival (EFS) as assessed by Investigator | Up to approximately 8 years
Percentage of participants who experience an adverse event (AE) | Up to approximately 60 weeks
Overall survival (OS) | Up to approximately 8 years
Health-Related Quality of Life (HR-QoL) score | Up to approximately 27-30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Jia, Study Chair — Tianjin Medical University Cancer Institute and Hospital; Jun Zhang, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No